CLINICAL TRIAL: NCT00360178
Title: An Open-label, Multicenter Study to Evaluate the Efficacy and Tolerability of a 4 Week Therapy With the Fixed Dose Combination of Valsartan 160 mg Plus HCTZ 25 mg in Hypertensive Patients Not Adequately Responding to a 4 Week Therapy With the Free Combination of an Angiotensin Receptor Blocker (Candesartan 32 mg) Plus HCTZ 25 mg
Brief Title: Efficacy and Safety of Valsartan Plus Hydrochlorothiazide in Fixed Dose Combination in Hypertensive Patients Not Controlled by the Free Combination of an Angiotensin Receptor Blocker Plus Hydrochlorothiazide
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVAH631BDE13
Record Dates: First submitted 2006-08-02; First posted 2006-08-04 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Hypertension
Keywords: hypertension; valsartan; amlodipine; hydrochlorothiazide
MeSH Terms: conditions — Hypertension | interventions — Valsartan; Hydrochlorothiazide; candesartan; Amlodipine

INTERVENTIONS:
Drug: Valsartan plus Hydrochlorothiazide
Drug: Candesartan plus Hydrochlorothiazide
Drug: Amlodipine

SUMMARY:
Recruiting in Germany only:

This study will evaluate the safety and efficacy of valsartan plus HCTZ in fixed dose combination in hypertensive patients not responding to treatment with the free combination of Candesartan plus HCTZ. In an optional extension patients with uncontrolled BP at the end of the core study can be treated with valsartan plus HCTZ in fixed dose combination plus amlodipine 5 mg for additional 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients (>=18 years)
2. Females must be either post-menopausal for one year, surgically sterile or using effective contraceptive methods (e.g. intra-uterine device, hormonal contraceptives).
3. Patients with moderate essential hypertension (WHO):

Exclusion Criteria:

1. Severe hypertension (WHO)
2. Pregnant or nursing women
3. Treated hypertensive patients with controlled hypertension under current therapy (MSDBP < 90 mmHg and MSSBP < 140 mmHg)
4. A history of cardiovascular disease, including angina pectoris, myocardial infarction, coronary artery bypass graft, percutaneous transluminal coronary angioplasty, transient ischemic attack, stroke, and heart failure NYHA II - IV

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2006-07; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Diastolic Blood Pressure (DBP) reduction by Valsartan + HCTZ in patients not adequately responding (i.e., DBP >= 90 mmHg) to 4 weeks of treatment with Candesartan + HCTZ in free combination
For optional extension: DBP reduction by Valsartan + HCTZ + Amlodipine in patients not adequately responding (i.e., DBP >= 90 mmHg and/or Systolic Blood Pressure (SBP) >= 140 mmHg) to 4 weeks of treatment with angiotensin receptor blockers + HCTZ

SECONDARY OUTCOMES:
SBP, pulse pressure, heart rate, normalization (DBP < 90 mmHg and/or SBP < 140 mmHg, resp.)and responder rate(DBP < 90 mmHg or reduction by at least 10 mmHg and/or SBP < 140 mmHg or reduction by at least 20 mmHg, rep)
Safety and tolerability
Compliance by pill count
For optional extension: SBP, pulse pressure, heart rate, normalization and responder rate as defined above

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceutical, Study Director — Sponsor GmbH
Locations (2):
- Investigative Centers, Germany
- Novartis Pharmaceuticals, Basel, Switzerland

REFERENCES:
- [Result] Schweizer J, Hilsmann U, Neumann G, Handrock R, Klebs S. Efficacy and safety of valsartan 160/HCTZ 25 mg in fixed combination in hypertensive patients not controlled by candesartan 32 mg plus HCTZ 25 mg in free combination. Curr Med Res Opin. 2007 Nov;23(11):2877-85. doi: 10.1185/030079907x242539. PMID 17922981